CLINICAL TRIAL: NCT02550821
Title: Comparison of Physical Activity Level Between Patients With Bronchiectasis and Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan CAKMAK, Research Assistant, Hacettepe University
Other Study IDs: GO 15/313
Record Dates: First submitted 2015-09-13; First posted 2015-09-16 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Bronchiectasis
Keywords: Physical activity levels; Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare physical activity levels between patients with bronchiectasis and healthy subjects.

We hypothesize that patients with bronchiectasis will have lower levels of physical activity, since physical activity levels is affected by reduced exercise tolerance, severity of disease and other disease related symptoms and conditions.

DETAILED DESCRIPTION:
Physical activity limitation in chronic respiratory diseases is caused by many factors including respiratory, hemodynamic, and peripheral muscle weakness. Bronchiectasis is characterized by irreversible widening of the medium-sized airways, with inflammation, chronic bacterial infection and destruction of the bronchial walls. In addition to pulmonary function worsening, extra pulmonary features such as reduced peripheral muscle endurance can be a significant physical problem which causing a decrease in physical activity levels.

Despite physical activity is considered to be essential for the management of chronic respiratory diseases, there is a lack of scientific study, which compares physical activity levels between patients with bronchiectasis and healthy subjects.

This study will assess physical activity level, exercise capacity, quality of life and peripheral muscle strength in patients with bronchiectasis compared to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of the Bronchiectasis Group:

1. Diagnosis of bronchiectasis
2. Being 18 years of age or older
3. Able and willing to complete the informed consent process.
4. Able to walk and co-operate

Exclusion Criteria:

Exclusion criteria of Bronchiectasis Group:

1. Unstable medical condition
2. To have severe neurological, orthopedic problems or severe heart failure.

The control group will consist of healthy subjects.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with bronchiectasis and healthy subjects.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of steps on accelerometer | Seven days
  Participants will wear an accelerometer (physical activity monitor) for seven consecutive days.
Energy expenditure on activity monitor | Seven days
  Total energy expenditure will be calculated using activity monitor for seven consecutive days
Exercise capacity using 6-minute walk test and incremental shuttle walk test | 8th day (after using device)
  6-minute walk test will be performed in a long, straight, enclosed corridor 30 meters in length. Patients are required to walk in their walking speed with standardized instructions. The distance walked by subjects during 6 minutes will be recorded.
  The incremental shuttle walk test will be performed in an enclosed corridor. Patients are required to walk back and forth, turning around two cones placed 9 meters apart making the shuttle distance 10 meters long. Patients will follow the rhythm dictated by the audio signal.
Physical activity level using International Physical Activity Questionnaire | 8th day
  Instrument to obtain internationally comparable data on health related physical activity This measure assesses the types of intensity of physical activity and sitting time in daily life and estimates total physical activity in MET-min/week and time spent sitting. It comprises open-ended questions surrounding individuals' last 7-day recall of physical activity.

SECONDARY OUTCOMES:
Shortness of breath using the Modified Medical Research Council Dyspnea Scale | 1st day (before using device)
  Scale is used to establish functional impairment due to dyspnea attributable to respiratory disease. The scoring ranges from 0 to 4. The higher scores indicate higher perception of dyspnea.
Quality of Life using St. George Respiratory Questionnaire | 1st day
  It measures the health impairment. The questionnaire consist of 50 items, 2 parts (3 components). The name of categories/domains were stated as follows: Part 1: Symptoms component (frequency&severity), Part 2: Activities that cause or are limited by breathlessness; Impact components (social functioning, psychological disturbances resulting from airways disease). The scores range from 0 to 100, with higher scores indicating more limitations.
Peripheral muscle strength test using a hand-held dynamometer | 8th day (after using device)
  Measurement of peripheral muscle strength
Maximal inspiratory and expiratory pressures measurement using a mouthpiece device | 8th day (after using device)
  Measurement of respiratory muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: ASLIHAN CAKMAK, Principal Investigator — Hacettepe University
Locations (1):
- Aslihan Cakmak, Ankara, Turkey (Türkiye)